CLINICAL TRIAL: NCT06630520
Title: Intraoperative Periarticular Injection May Improve Postoperative Pain Scores and Reduce Opioid Consumption in Arthroscopic Anterior Cruciate Ligament Reconstruction Surgery
Brief Title: Intraoperative Periarticular Injection in Arthroscopic Anterior Cruciate Ligament Reconstruction Surgery
Acronym: PAI in ACLR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, En-Rung Chiang, Division Director, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-05-004B
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2022-02

CONDITIONS: Anterior Cruciate Ligament (ACL) Tear; Arthroscopic Anterior Cruciate Ligament Reconstruction
Keywords: periarticular injection; morphine consumption; pain control
MeSH Terms: conditions — Lacerations; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Periarticular injection (Active Comparator)
  Interventions: Combination Product: Periarticular injection
- Control group (No Intervention)

INTERVENTIONS:
Combination Product: Periarticular injection — A 50ml periarticular injection was introduced intraoperatively before the time of closing. The injection contained 150mg bupivacaine (3mg/mL), 60mg ketorolac(1.2mg/mL) and 1mg morphine.
  Before wound closure, periarticular cocktail was injected around the knee joint including the adductor canal from the hamstring harvest side in PAI group. All patients had oral paracetamol 500mg, 4 times/day and diclofenac 75mg, 1 times/day after surgery.
  Arms: Periarticular injection

SUMMARY:
In this prospective, assessor-blinded, single-surgeon clinical trial, the goal was to validate the efficacy of PAI in aACLR surgery with a reduced opioid dose, while achieving similar pain relief with few adverse events. 300 patients who had undergone aACLR were randomly allocated to receive either a PAI or nPAI group. The primary outcome parameters were visual analogue scale (VAS) scores and cumulative morphine dose, through time. Secondary outcome parameters included drug-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients 18 years or older who had undergone a-ACLR with or without meniscus procedure for anterolateral instability of the knee; 2) agree to participate in this study and to be randomly allocated to either or peri-articular injection protocol and have signed an informed consent.

Exclusion Criteria:

* 1) patients with other concomitant injuries such as other ligamentous injury or fracture; 2) Allergy to any of the medication used in either protocol; 3) patient with history of the chronic pain 4) preoperative chronic opioid-dependent patients (exceeding 50 mg oral morphine equivalence per day at time of recruitment); 5) refuse to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
VAS scores | at different time points (postoperative 4,8,24-hour, before discharge) after surgery

SECONDARY OUTCOMES:
cumulative morphine consumption (mg) | at post-operative 4, 8, 24-hour and before discharge

OTHER OUTCOMES:
drug related adverse events | within postoperative 2 weeks
overall satisfaction scale (0-100 points) | at postoperative 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Concerning the patient's privacy